CLINICAL TRIAL: NCT00445809
Title: EValuation Of NGAL in Early and eVolving Acute kidnEy Injury
Brief Title: Evaluation of Neutrophil Gelatinase-associated Lipocalin (NGAL) in Early and Evolving Acute Kidney Injury
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Kyle Fortner, CRA, Biosite, Incorporated a subsidiary of Inverness Medical Innovations
Other Study IDs: BSTE-0401
Record Dates: First submitted 2007-02-15; First posted 2007-03-09 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Kidney Failure, Acute
Keywords: Kidney; Renal; Cardiac Surgery with bypass; Cardiovascular surgery with cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples (3 10ml, 7 5ml) at ten timepoints over 5 days.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: High Risk population for developing AKI during/after CABG surgery.
- 2: Medium Risk population for developing AKI during/after CABG surgery.

SUMMARY:
Some patients who undergo cardiovascular surgery requiring cardiopulmonary bypass will develop a kidney injury following their surgery. The purpose of this study is to take a blood sample from patients before they have this type of surgery and then at nine time points after their surgery to test their plasma for a biomarker called NGAL and compare the NGAL levels to their creatinine levels. We hypothesize that NGAL is an earlier marker for kidney injury than creatinine.

DETAILED DESCRIPTION:
Approximately 350 adults scheduled to undergo cardiac surgery involving the use of cardiopulmonary bypass will be enrolled. Blood samples will be obtained from all patients in the study for future measurement of both plasma NGAL and plasma creatinine levels in the same sample at each of nine time points.

Blood samples for later assessment using the Triage NGAL Test will be processed to plasma at the clinical site, frozen and shipped to Biosite for storage. Testing with the Triage NGAL Test will be conducted at Biosite by trained laboratory personnel. The results of these assessments will be blinded to the medical team during the study and will not impact the medical management of the patient.

The medical team caring for each study patient should obtain clinical laboratory tests per their usual post-operative routine and manage the patient accordingly. Any serum creatinine measurements obtained by the site as part of this routine care both pre-operatively and through Day 10 post-operatively will be recorded as well as any additional post-operative renal insults, the development of oliguria, the need for a nephrology consultation, initiation of dialysis and mortality will also be recorded through Day 10.

ELIGIBILITY:
4.2.1 Inclusion Criteria

1. Male or female scheduled for cardiovascular surgery (other than cardiac transplant) requiring cardiopulmonary bypass
2. 18 years of age or older

i. The first approximately 150 to200 patients enrolled must have:

• A Prediction of Acute Renal Failure Score ≥ 5 (see Reference 18 and Appendix B)

ii. The subsequent patients enrolled must have one or more of the following risk factors for post-bypass renal injury:

* Age > 70;
* Pre-operative creatinine > 1.4 mg/dL;
* NYHA Class 3 or 4 heart failure or left ventricular ejection fraction < 35%;
* Insulin-dependent diabetes mellitus;
* Undergoing cardiac valve surgery;
* History of previous cardiac surgery.

Exclusion Criteria:

* Age < 18 years
* Inability to obtain Informed Consent from patient or representative
* Prisoners or other institutionalized or vulnerable individuals
* Participation in an interventional clinical study within the previous 30 days
* History of previous renal transplantation
* Stage 5 chronic kidney disease (estimated GRF<15 mL/min/1.73m2) (See Appendix C)
* Known or suspected ongoing pre-operative acute renal failure due to any cause, including pre-renal, intrinsic renal or post-renal (obstructive) etiologies (as evidenced by increasing serum creatinines or oliguria pre-operatively)
* Already receiving dialysis, in imminent need of dialysis or considered highly likely to need dialysis in the immediate post-operative period for fluid management
* Any known or suspected renal ischemic insult(such as cardiac arrest)or nephrotoxic insult(other than intravascular contrast procedure) during the 48 hours prior to surgery
* Known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV)infection, hepatitis B virus (HBV) infection or other infectious hepatitis
* Pre-operative hematocrit <25%, recent blood transfusions have been administered to maintain hematocrit >25% or any other contraindication to obtaining the study-specified blood samples
* Undergoing cardiac transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CABG Surgery that are thought to have a risk of developing AKI during/after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil Paganini, MD, Principal Investigator — The Cleveland Clinic
Locations (11):
- United States (10):
  - St. Anthony's Central Hospital, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Maine Medical Center, Portland, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Peters Healthcare, Albany, New York
  - New York Methodist, Brooklyn, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Houston, Houston, Texas
- University of British Columbia, Vancouver, British Columbia, Canada